CLINICAL TRIAL: NCT00057811
Title: A Pilot Study To Determine The Toxicity Of The Addition Of Rituximab To The Induction And Consolidation Phases And The Addition Of Rasburicase To The Reduction Phase In Children With Newly Diagnosed Advanced B-Cell Leukemia/Lymphoma Treated With LMB/FAB Therapy
Brief Title: Rituximab, Rasburicase, and Combination Chemotherapy in Treating Young Patients With Newly Diagnosed Advanced B-Cell Leukemia or Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANHL01P1; NCI-2009-00405 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ANHL01P1 (Other: Children's Oncology Group); CDR0000271941 (Other: Clinical Trials.gov); U10CA098543 (NIH)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Childhood Burkitt Lymphoma; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Stage I Childhood Large Cell Lymphoma; Stage I Childhood Small Noncleaved Cell Lymphoma; Stage II Childhood Large Cell Lymphoma; Stage II Childhood Small Noncleaved Cell Lymphoma; Stage III Childhood Large Cell Lymphoma; Stage III Childhood Small Noncleaved Cell Lymphoma; Stage IV Childhood Large Cell Lymphoma; Stage IV Childhood Small Noncleaved Cell Lymphoma; Untreated Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating | interventions — Doxorubicin; Cyclophosphamide; Methotrexate; merphos; rasburicase; Peplomycin; Urate Oxidase; Leucovorin; Prednisone; Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; Filgrastim; Granulocyte Colony-Stimulating Factor; Rituximab; Cytarabine; Etoposide; Vincristine; Hydrocortisone; hydrocortisone hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group B (chemotherapy, protective therapy, monoclonal antib.) (Experimental): Therapies given IV, IT, orally, or SC. Please see treatment outline. See Detailed Description.
  Interventions: Drug: doxorubicin hydrochloride; Drug: cyclophosphamide; Drug: methotrexate; Drug: rasburicase; Drug: leucovorin calcium; Drug: prednisone; Drug: methylprednisolone; Biological: filgrastim; Biological: rituximab; Drug: cytarabine; Drug: vincristine sulfate; Drug: hydrocortisone sodium succinate; Other: laboratory biomarker analysis
- Group C (Chemotherapy, monoclonal antibody therapy) (Experimental): Therapies given IV, IT, orally, or subcutaneously (same as FAB B with the addition of etoposide and high-dose methotrexate). See Detailed Description.
  Interventions: Drug: doxorubicin hydrochloride; Drug: cyclophosphamide; Drug: methotrexate; Drug: leucovorin calcium; Drug: prednisone; Drug: methylprednisolone; Biological: filgrastim; Biological: rituximab; Drug: cytarabine; Drug: etoposide; Drug: vincristine sulfate; Drug: hydrocortisone sodium succinate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Given IV, IT, or orally
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: methotrexate — Given IV or IT
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: rasburicase — Given IV
  Other Names: Elitek; NK-631; recombinant urate oxidase
  Arms: Group B (chemotherapy, protective therapy, monoclonal antib.)
Drug: leucovorin calcium — Given IV or orally
  Other Names: CF; CFR; LV
Drug: prednisone — Given IV or orally
  Other Names: DeCortin; Deltra
Drug: methylprednisolone — Given IV or orally
  Other Names: Depo-Medrol; Medrol; MePRDL; Solu-Medrol; Wyacort
Biological: filgrastim — Given subcutaneously
  Other Names: G-CSF; Neupogen
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: cytarabine — Given IT
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
  Arms: Group C (Chemotherapy, monoclonal antibody therapy)
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: hydrocortisone sodium succinate — Given IT
  Other Names: Sodium hydrocortisone succinate; Solu-Cortef; Solu-Glyc
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of combining rituximab and rasburicase with combination chemotherapy in treating young patients who have newly diagnosed advanced B-cell leukemia or lymphoma. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug with rituximab may kill more cancer cells. Chemoprotective drugs such as rasburicase may protect kidney cells from the side effects of chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the toxicity of the addition of rituximab to induction chemotherapy comprising vincristine, methylprednisolone, methotrexate, leucovorin calcium, cyclophosphamide, and doxorubicin (COPADM) [COMRAP] and to consolidation chemotherapy in children with newly diagnosed FAB prognostic group B or group C leukemia or lymphoma treated with LMB/FAB therapy.

II. Determine the toxicity of the addition of rasburicase to the reduction phase comprising cyclophosphamide, vincristine, prednisone or methylprednisolone, methotrexate, and leucovorin calcium (COP-R) in these patients.

III. Determine the incidence of tumor lysis syndrome, renal complications, and the use of assisted renal support (i.e., dialysis or hemofiltration) during the COP-R reduction phase and the first induction phase of COPADM or COMRAP in these patients.

IV. Determine the response rate of patients treated with COMRAP incorporated into LMB/FAB therapy.

V. Assess minimal residual disease in patients before and during COMRAP therapy incorporated into LMB/FAB therapy.

OUTLINE: This is a multicenter study. Patients are stratified according to FAB prognostic group (B vs C) and treated by group classification.

FAB GROUP B

TREATMENT I (first 6 patients):

REDUCTION THERAPY: Patients receive the COP-R regimen comprising cyclophosphamide IV over 15 minutes, vincristine IV, and methotrexate and hydrocortisone intrathecally (IT) on day 0; rasburicase* IV over 30 minutes every 12 hours on days 0 and 1 and then once daily on days 2-4 (patients exhibiting hyperuricemia and clinical suspicion of B-cell non-Hodgkin's lymphoma or B-cell acute lymphocytic leukemia also receive rasburicase on days -3, -2, and -1); leucovorin calcium IV or orally every 12 hours on days 1 and 3; and prednisone (PRED) or methylprednisolone (MePRDL) IV (or orally) on days 0-6. Patients too critical to proceed may receive another course of reduction therapy.

NOTE: *Patients with G6PD deficiency do not receive rasburicase during reduction therapy.

INDUCTION THERAPY: Patients with less than 20% tumor reduction follow the group C induction phase (described below). Patients with at least 20% tumor reduction receive 1 course of the COPADM regimen: vincristine IV and methotrexate IV over 4 hours on day 0; PRED or MePRDL IV (or orally) on days 0-7; leucovorin calcium IV or orally every 6 hours for 12 doses on days 1-3; doxorubicin IV over 30-60 minutes on day 1; cyclophosphamide IV over 15 minutes every 12 hours on days 1-3; methotrexate IT and hydrocortisone IT on days 1 and 5; and filgrastim (G-CSF) subcutaneously (SC) beginning on day 6 and continuing until blood counts recover.

Patients receive the second part of induction therapy when peripheral blood counts have recovered but no fewer than 16 days after the first part of induction therapy. Patients receive 1 course of the COMRAP regimen comprising rituximab IV on days -2 and 0 with COPADM as in the first part of induction therapy.

CONSOLIDATION THERAPY: Patients receive the CYM-RM regimen comprising rituximab IV and methotrexate IV over 4 hours on day 0; leucovorin calcium IV or orally every 6 hours for 12 doses on days 1-3; cytarabine IV over 24 hours daily on days 1-5; hydrocortisone IT on days 1 and 6; methotrexate IT on day 1; and cytarabine IT on day 6.

After full recovery from consolidation therapy, patients with any residual masses undergo surgical excision or biopsy. Patients with histology positive for tumor (even if completely resected) proceed to Group C consolidation therapy (described below). Patients with histology negative for tumor proceed to Group B maintenance therapy.

MAINTENANCE THERAPY: Patients receive the COPADM regimen comprising vincristine IV and methotrexate IV over 4 hours on day 0; PRED or MePRDL IV (or orally) on days 0-7; doxorubicin IV over 30-60 minutes, and cyclophosphamide IV over 30 minutes on days 1 and 2; methotrexate IT and hydrocortisone IT on day 1; and leucovorin calcium IV or orally every 6 hours on days 1-3 (12 doses).

TREATMENT II (44 patients):

REDUCTION THERAPY: Patients receive the COP-R regimen as in treatment I.

INDUCTION THERAPY: Patients receive 2 courses of the COMRAP regimen as in the second induction of treatment I.

CONSOLIDATION THERAPY: Patients receive the CYM-RM regimen as in treatment I.

MAINTENANCE THERAPY: Patients receive the COPADM regimen as in treatment I.

FAB GROUP C:

TREATMENT I (first 3 patients):

REDUCTION THERAPY: Patients receive the COP-R regimen as in group B treatment I, with the addition of triple intrathecal therapy (TIT) comprising methotrexate, hydrocortisone, and cytarabine on days 0, 2, and 4.

INDUCTION THERAPY: Patients receive 2 courses of the COPADM regimen as in group B treatment I, with the addition of TIT on days 1, 3, and 5. Patients in group C who have biopsy-proven disease after induction therapy are off protocol therapy and treated at the discretion of the investigator.

CONSOLIDATION THERAPY:

CNS-POSITIVE DISEASE: Patients receive 2 courses of the CYVE-RM regimen comprising rituximab IV and methotrexate and hydrocortisone IT on day 0; cytarabine IV over 12 hours on days 0-4; high-dose cytarabine IV over 3 hours and etoposide IV over 2 hours on days 1-4; and G-CSF SC on days 6-20. During the first course, patients also receive HD-MTX IV over 4 hours on day 17; TIT on day 18; and leucovorin calcium IV or orally every 6 hours on days 18-21 (12 doses).

CNS-NEGATIVE DISEASE: Patients receive the CYVE-RM regimen without intrathecal therapy, HD-MTX, or leucovorin calcium.

After full recovery from consolidation therapy, patients with any residual masses undergo surgical excision or biopsy. Patients who do not achieve complete remission after consolidation therapy are considered treatment failures.

MAINTENANCE THERAPY (each course lasts 28 days):

COURSE M1: Patients receive vincristine IV and high-dose methotrexate IV over 4 hours on day 0; PRED or MePRDL IV (or orally) on days 0-7; doxorubicin IV over 30-60 minutes and TIT on day 1; cyclophosphamide IV over 30 minutes on days 1 and 2; and leucovorin calcium IV or orally every 6 hours on days 1-4 (12 doses).

COURSE M2: Patients receive etoposide IV over 90 minutes on days 0-2 and cytarabine SC every 12 hours on days 0-4.

COURSE M3: Patients receive vincristine IV on day 0; cyclophosphamide IV over 30 minutes on days 0 and 1; PRED or MePRDL IV (or orally) twice daily on days 0-7; and doxorubicin IV over 30-60 minutes on day 0 (after first dose of cyclophosphamide).

COURSE M4: Patients receive etoposide and cytarabine as in course M2.

TREATMENT II (37 patients):

REDUCTION THERAPY: Patients receive 2 courses of the COP-R regimen as in group C treatment I.

INDUCTION THERAPY: Patients receive the COMRAP regimen comprising rituximab IV, vincristine IV, and HD-MTX IV over 4 hours on day 0; PRED or MePRDL IV (or orally) on days 0-7; leucovorin calcium IV or orally and cyclophosphamide IV over 15 minutes on days 1-3; doxorubicin IV over 30-60 minutes on day 1; TIT on days 1, 3, and 5; and G-CSF SC on days 6-20.

CONSOLIDATION THERAPY: CNS-positive disease: Patients receive the CYVE-RM regimen plus HD-MTX as in group C treatment I. Patients then receive CYVE-RM for a second course.

CNS-NEGATIVE DISEASE: Patients receive CYVE-RM regimen as in group C treatment I.

MAINTENANCE THERAPY: Patients receive maintenance therapy as in group C treatment I.

Patients are followed every 3-6 months for 1 year and then every 6 months for up to 5 years

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed mature B-lineage (CD20-positive) leukemia or lymphoma by the REAL classification of 1 of the following subtypes:

  * Diffuse large cell lymphoma
  * Burkitt's lymphoma
  * High-grade B-cell lymphoma (Burkitt-like)
* No B-cell anaplastic large cell Ki-1 positive lymphomas and B-lymphoblastic lymphomas
* One of the following FAB prognostic groups:

  * Group B (intermediate risk)
  * Group C (high risk)

    * Bone marrow involvement with at least 25% blasts and/or CNS involvement meeting 1 or more of the following criteria:

      * Any L3 blasts in cerebrospinal fluid
      * Cranial nerve palsy (if not explained by extracranial tumor)
      * Clinical spinal cord compression
      * Isolated intracerebral mass
      * Parameningeal extension (cranial and/or spinal)
* Hepatitis B status known
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* No known history of congenital immune deficiency and/or laboratory evidence of acquired immune deficiency
* No known G6PD deficiency (if receiving rasburicase)
* No prior malignancies treated with systemic chemotherapy with alkylator or anthracycline therapy
* No prior chemotherapy
* At least 1 week since prior steroids except emergency steroids initiated within 72 hours of study entry
* No prior radiotherapy except emergency radiotherapy initiated within 72 hours of study entry
* No concurrent radiotherapy
* No prior solid organ transplantation

Ages: 1 Year to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2004-06; Primary Completion 2009-10 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Cairo, MD CCRP, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States

REFERENCES:
- [Background] Shiramizu B, Goldman S, Kusao I, Agsalda M, Lynch J, Smith L, Harrison L, Morris E, Gross TG, Sanger W, Perkins S, Cairo MS. Minimal disease assessment in the treatment of children and adolescents with intermediate-risk (Stage III/IV) B-cell non-Hodgkin lymphoma: a children's oncology group report. Br J Haematol. 2011 Jun;153(6):758-63. doi: 10.1111/j.1365-2141.2011.08681.x. Epub 2011 Apr 18. PMID 21496005
- [Derived] Frazer JK, Li KJ, Galardy PJ, Perkins SL, Auperin A, Anderson JR, Pinkerton R, Buxton A, Gross TG, Michon J, Leverger G, Weinstein HJ, Harrison L, Shiramizu B, Barth MJ, Goldman SC, Patte C, Cairo MS. Excellent outcomes in children and adolescents with CNS+ Burkitt lymphoma or other mature B-NHL using only intrathecal and systemic chemoimmunotherapy: results from FAB/LMB96 and COG ANHL01P1. Br J Haematol. 2019 Apr;185(2):374-377. doi: 10.1111/bjh.15520. Epub 2018 Aug 16. No abstract available. PMID 30117142

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group B (Chemotherapy, Protective Therapy, Monoclonal Antib.) | Group C (Chemotherapy, Monoclonal Antibody Therapy)
Started | 51 | 46
Completed | 41 | 34
Not Completed | 10 | 12
Not completed — Lack of Efficacy | 1 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Ineligible | 4 | 2
Not completed — Inevaluable | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group B (Chemotherapy, Protective Therapy, Monoclonal Antib.) | Group C (Chemotherapy, Monoclonal Antibody Therapy) | Total
Number analyzed (Participants) | 51 | 46 | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 49 | 44 | 93
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 4575 [2497 to 5638] | 3132 [1940 to 4419] | 3853.5 [2218.5 to 5028.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 41 | 37 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 19
  Not Hispanic or Latino | 39 | 36 | 75
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 40 | 34 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 47 | 38 | 85
  Australia | 1 | 3 | 4
  Canada | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Grade ≥ 3 Stomatitis
Description: The incidence of grade ≥ 3 stomatitis. Grade 3 stomatitis: Confluent ulcerations or pseudomembranes; bleeding with minor trauma. Grade 4 stomatitis: Tissue necrosis; Significant spontaneous bleeding; life-threatening consequences
Time Frame: Up to 1 year
Population: Population analyzed includes eligible patients (Group B:46; Group C: 42). Three additional patients (Group B:1; Group C:2) have been excluded as inevaluable per the study chair.
Measure: Number; unit: participants
Arm/Group | Group B (Chemotherapy, Protective Therapy, Monoclonal Antib.) | Group C (Chemotherapy, Monoclonal Antibody Therapy)
Number analyzed (Participants) | 45 | 40
participants
  Incidence of grade ≥ 3 stomatitis | 4 | 6
  No incidence of grade ≥ 3 stomatitis | 41 | 34

2. Primary Outcome: Response Rate
Description: Response includes both complete and partial responses. Per protocol, complete Response is defined as the complete disappearance of all clinical evidence of disease by physical examination, by imaging studies, by bone marrow biopsy (where indicated), by CNS evaluation (where indicated) and by biopsy where there is a residual abnormality on an imaging study. Bone marrow must contain <5% blasts. CSF WBC must be <5/μL with no blasts or lymphomatous cells present. Partial response is defined as: at least a 50% reduction in the size of all measurable tumor areas. Each site is to be defined by the product of the maximum length, width and depth (3 dimensions). No lesion may progress. No new lesion may appear. Bone marrow must contain <5% blasts. CSF WBC must be <5/μL with no blasts or lymphomatous cells present..
Time Frame: Up to 5 years
Population: Population analyzed includes eligible patients considered evaluable for response (with measurable disease at on study and adequate assessment of response).
Measure: Number (95% Confidence Interval); unit: percentage of participants analyzed
Arm/Group | Group B (Chemotherapy, Protective Therapy, Monoclonal Antib.) | Group C (Chemotherapy, Monoclonal Antibody Therapy)
Number analyzed (Participants) | 32 | 23
percentage of participants analyzed | 88 [71 to 96] | 83 [61 to 95]

3. Primary Outcome: Minimal Residual Disease
Description: The presence or absence of tumor cells at the end of induction assessed by studying tissue and/or blood/marrow. Details of methods and criteria used can be found in Shiramizu at al. BJH 153:758-763, 2011 (full citation in the citation section).
Time Frame: Not Provided
Population: Population analyzed included patients submitting samples for minimal disease assay at end induction
Measure: Number (95% Confidence Interval); unit: percentage of samples analyzed
Arm/Group | Group B (Chemotherapy, Protective Therapy, Monoclonal Antib.) | Group C (Chemotherapy, Monoclonal Antibody Therapy)
Number analyzed (Participants) | 32 | 10
percentage of samples analyzed | 22 [11 to 40] | 70 [35 to 93]

4. Primary Outcome: Toxic Death
Description: Implementation of the toxic death rate stopping rule, a death must be possibly, probably or definitely attributable to Rituximab and/or chemotherapy to be considered a toxic death.
Time Frame: Up to 1 year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Group B (Chemotherapy, Protective Therapy, Monoclonal Antib.) | Group C (Chemotherapy, Monoclonal Antibody Therapy)
Number analyzed (Participants) | 45 | 40
participants
  Toxic death | 0 | 2
  No toxic death | 45 | 38

ADVERSE EVENTS:
Description: For Group B, 46 participants are reported for adverse events as 5 patients were declared ineligible. For Group C, 42 participants are reported for adverse events as 4 patients were declared ineligible.
Arm/Group | Group B (Chemotherapy, Protective Therapy, Monoclonal Antib.) | Group C (Chemotherapy, Monoclonal Antibody Therapy)
Serious Adverse Events (participants affected / at risk) | 2/46 | 6/42
Other Adverse Events (participants affected / at risk) | 32/46 | 35/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group B (Chemotherapy, Protective Therapy, Monoclonal Antib.) (N=46) | Group C (Chemotherapy, Monoclonal Antibody Therapy) (N=42)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 6 (6)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 3 (3)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group B (Chemotherapy, Protective Therapy, Monoclonal Antib.) (N=46) | Group C (Chemotherapy, Monoclonal Antibody Therapy) (N=42)
Anemia (Blood and lymphatic system disorders) | 32 (32) | 32 (32)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 18 (18) | 22 (22)
Asystole (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 2 (2)
Mobitz type I (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 2 (2)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 2 (2) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 11 (11)
Anal mucositis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 13 (13)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 19 (19) | 18 (18)
Nausea (Gastrointestinal disorders) | 10 (10) | 15 (15)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Oral pain (Gastrointestinal disorders) | 3 (3) | 7 (7)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 8 (8) | 13 (13)
Chills (General disorders) | 2 (2) | 2 (2)
Edema limbs (General disorders) | 0 (0) | 4 (4)
Fatigue (General disorders) | 1 (1) | 7 (7)
Fever (General disorders) | 4 (4) | 11 (11)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 7 (7) | 5 (5)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 5 (5) | 2 (2)
Anaphylaxis (Immune system disorders) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 5 (5)
Enterocolitis infectious (Infections and infestations) | 5 (5) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 16 (16) | 23 (23)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Small intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Venous injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 27 (27) | 25 (25)
Alkaline phosphatase increased (Investigations) | 5 (5) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 16 (16) | 21 (21)
Blood bilirubin increased (Investigations) | 1 (1) | 13 (13)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 6 (6) | 8 (8)
Fibrinogen decreased (Investigations) | 0 (0) | 1 (1)
GGT increased (Investigations) | 0 (0) | 8 (8)
INR increased (Investigations) | 1 (1) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 5 (5)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 9 (9) | 9 (9)
Neutrophil count decreased (Investigations) | 31 (31) | 35 (35)
Platelet count decreased (Investigations) | 29 (29) | 34 (34)
Serum amylase increased (Investigations) | 0 (0) | 3 (3)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 3 (3) | 6 (6)
White blood cell decreased (Investigations) | 31 (31) | 29 (29)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 12 (12)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 20 (20) | 18 (18)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 (13) | 18 (18)
Hypocalcemia (Metabolism and nutrition disorders) | 16 (16) | 20 (20)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 17 (17) | 23 (23)
Hypomagnesemia (Metabolism and nutrition disorders) | 10 (10) | 9 (9)
Hyponatremia (Metabolism and nutrition disorders) | 16 (16) | 16 (16)
Hypophosphatemia (Metabolism and nutrition disorders) | 14 (14) | 11 (11)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Abducens nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 9 (9) | 8 (8)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 3 (3) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Body odor (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 12 (12)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 10 (10)
Hypotension (Vascular disorders) | 2 (2) | 9 (9)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.